CLINICAL TRIAL: NCT05590182
Title: Randomized-Controlled Study to Evaluate the Diagnostic Quality and Safety of Automated Carbon Dioxide Angiography (ACDA) With a Robot-supported Angiography System in Combination With a CO2-Injector System in Patients With Peripheral Arterial Occlusive Disease
Brief Title: CO2-Angiography-Study to Evaluate Diagnostic and Safety to Patients With Peripher Arterial Stenotic or Occlusive Disease.
Acronym: ACDA-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: AngioDroid s.r.l., Bologna (Italy) (Unknown)
Responsible Party: Principal Investigator, René Aschenbach, Head Interventional Radiology,, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 5168-05/17
Record Dates: First submitted 2017-07-17; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: CO2; angiography; peripheral occlusion disease; contrast medium; carbon dioxid enhanced angiography
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — Angiography

STUDY DESIGN:
Intervention Model Description: The randomization that allocates the patient either in the study arm (CO2) or in the control arm (iodine-CM) will occur right before angiography. Stenosis graduation and length will be measured after diagnostic angiography and before intervention. The interventional angiography will be conducted with the opposed contrast media used for diagnostic angiography. If contrast media containing iodine was used for diagnostic angiography, CO2 must be used for interventional angiography and if CO2 was applied for diagnostic angiography, contrast media containing iodine must be used for interventional angiography. The calculated values through the software-quantification-tool, including also a final sequence of the distal outflow with the same contrast media used during intervention, are be compared and statistically analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO2 first/ iodine CM second (Active Comparator): CO2-enhanced angiography
  Interventions: Device: Angiography
- iodine CM first/ CO2 second (Active Comparator): iodine contrast media-enhanced angiography
  Interventions: Device: Angiography

INTERVENTIONS:
Device: Angiography — Randomization either in the study arm (CO2) or in the control arm (iodine-CM) occurs right before angiography. Stenosis graduation and length are measured after diagnostic angiography and before intervention. The calculated values through the software-quantification-tool, including also a final sequence of the distal outflow with the same contrast media used during intervention, are be compared and statistically analyzed.
  A pain protocol to the current pain-situation is led by the present medical-laboratory assistant after administration of CO2 and iodine-CM during intervention.

SUMMARY:
This randomized study focuses on the diagnostic quality and safety of CO2 application as contrast medium through an innovative injector of AngioDroid in angiography interventions in patients with peripheral arterial occlusive diseases.

DETAILED DESCRIPTION:
CO2-angiography was used as an intra-arterial contrast agent since the 1970s particularly in patients who were hypersensitive to iodinated contrast material or whose renal function was compromised. It is in fact an effective and low-risk alternative to iodine-enhanced conventional angiography because it is not associated with nephrotoxicity or allergic reactions. The image quality influencing the diagnostic validity seems to be a restriction. Now, with the availability of high-resolution DSA and a reliable gas delivery system, CO2 angiography is more and more widely used for vascular imaging and endovascular procedures. Our study will specifically examine the image quality and safety of carbon dioxide gas as intra-arterial contrast agent using the innovative Artis Zeego Q angiography-system of Siemens Healthineers with the automated CO2-injection system of Angiodroid.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Male, female
* Patients with indication for percutaneous transluminal angioplasty of iliacal- or femoropopliteal arteries

Exclusion Criteria:

* Children and adolescents < 18 years
* Diagnostic angiography, CT- or MRI-angiography during the past 3 months
* Patients with reduced renal function (S-creatinine > 1,2 mg/dl)
* Incapacitated patients
* Severe COPD
* Known atrium- or ventricular septal defect with right-left-shunt
* Current participation in other interventional studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Degree of stenosis | during intervention
  Calculation of maximum grade of stenosis

SECONDARY OUTCOMES:
Image quality | 2 weeks
  Image quality assessed by blinded radiologists who did not perform the angiographic intervention.
occurence of adverse events | 24 hours
  Complications documted within 24 hours and pain scale during intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Teichgräber, Prof. Dr. med., Principal Investigator — University Hospital Jena, Radiology Department, Germany
Locations (1):
- University Hospital, Jena, Thuringia, Germany